CLINICAL TRIAL: NCT00563654
Title: Randomized Trial Comparing Alfuzosin GITS 10 mg Daily With Placebo on the Successful Rate of Trial Without Catheter in Patients With Acute Urinary Retention With Long Term Follow up
Brief Title: Randomized Trial Comparing Alfuzosin GITS 10 mg Daily With Placebo for Trial Without Catheter in Acute Urinary Retention With Long Term Follow up
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2005.332; HARECCTR0500048
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Prostatic Hyperplasia; Urinary Retention; Acute Disease
Keywords: Benign Prostatic Hyperplasia (BPH); Acute Retention of Urine (AUR)
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Retention; Acute Disease | interventions — alfuzosin

INTERVENTIONS:
Drug: Alfuzosin GITS (Xatral XL)

SUMMARY:
The purpose of the study is to compare alfuzosin GITS once daily versus placebo in achieving a successful TWOC after AUR due to BPH, among Chinese males in Hong Kong, and in delaying or avoiding a TURP.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 or above
* Admitted for AUR due to BPH with PVR of 500 ml or more

Exclusion Criteria:

* Previous history of TURP
* Use of alpha blockers within recent 8 months
* Renal impairment (serum creatinine >140 umol/l)
* Poor premorbid state

Min Age: 50 Years | Sex: Male
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-10; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Successful rate of Trial Without Catheter (TWOC) at phase 1 | At discharge after TWOC (at the end phase one)
Late failure of TWOC of, which is defined as recurrent of AUR or the need of invasive therapy among those who are successful in TWOC in phase 1 | From the end of phase one to eight months after successful TWOC (the end of phase 2)

SECONDARY OUTCOMES:
Proportion of subjects with hypotension or symptoms related to hypotension after administration of treatment drug for TWOC | From the time of treatment drug administration to the end of phase 1
Peak flow rate (Qmax), voided volume (Vcomp) and post-voided residue volume (PVR) | At the end of phase I (discharge after TWOC) and at the end of phase 2

CONTACTS AND LOCATIONS:
Overall Officials: Chi Wai Cheng, Dr, Principal Investigator — Department of Surgery, Division of Urology, North District Hospital
Locations (1):
- North District Hospital, Hong Kong, China